CLINICAL TRIAL: NCT01775748
Title: Effect Of Concord Grape Juice On Endothelial Function In Obese And Overweight Individuals Over Age 50
Brief Title: Effect of Concord Grape Juice on Endothelial Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: Welch's, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: H-31937
Record Dates: First submitted 2013-01-23; First posted 2013-01-25 (Estimated); Last update posted 2018-02-12 (Actual); Status verified 2018-02

CONDITIONS: Obesity; Overweight
Keywords: Grape juice
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active First (Other): Active Concord Grape Juice 12 oz per day Placebo Grape Juice 12 oz per day
  Interventions: Other: Active Concord Grape Juice 12 oz per day; Other: Placebo Grape Juice 12 oz per day
- Placebo First (Other): Placebo Grape Juice 12 oz per day Active Concord Grape Juice 12 oz per day
  Interventions: Other: Active Concord Grape Juice 12 oz per day; Other: Placebo Grape Juice 12 oz per day

INTERVENTIONS:
Other: Active Concord Grape Juice 12 oz per day — Grape Juice 12 oz per day
Other: Placebo Grape Juice 12 oz per day — Placebo Grape Juice 12 oz per day

SUMMARY:
The study will compare Concord grape juice to a beverage that contains no grape flavonoids, but has a similar appearance and taste (placebo juice). A total of 60 overweight and obese participants over age 50 will be enrolled. Each participant will drink each beverage for 4 weeks with a 2-week rest period between two beverage consumption periods. The order of beverages (grape juice first or placebo juice first) will be randomized. The investigators will use ultrasound to measure brachial artery flow-mediated dilation, a measure of endothelial vasodilator function. The investigators will also collect blood samples to further assess the cardiovascular effects of grape juice.

The aim of the study is to determine whether Concord grape juice improves endothelial function in patients at risk who do not have cardiovascular disease and may provide information that would guide dietary recommendations. The results may also be used by the sponsor to substantiate claims and labeling of their product.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index ≥ 25 and < 40 kg/m2
* Age ≥ 50 years
* Otherwise healthy

Exclusion Criteria:

* Clinical diagnosis of atherosclerotic vascular disease.
* Clinical history of diabetes mellitus or fasting glucose ≥126 mg/dl
* Uncontrolled hypertension
* Treatment with an investigational new drug within the last 30 days
* Clinical history of other major illness including end-stage cancer, renal failure, hepatic failure, or other conditions that in the opinion of the principal investigator make the study inappropriate
* Psychological illness or condition such as to interfere with the subject's ability to understand the requirements of the study
* Use of Vitamin E, Vitamin C, beta carotene, lipoic acid, or other food or herbal supplements within 1 month of enrollment. Subjects taking multivitamins or other forms of vitamin E and C in doses that do not exceed two times the recommended daily allowance will not be excluded
* Extreme dietary habits (i.e. Atkins, very high protein/low carbohydrate, or vegan diet

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2014-03-19 (Actual); Study Completion 2014-03-19 (Actual)

PRIMARY OUTCOMES:
Brachial artery flow mediated dilation | 4 weeks
  Endothelial function will be assessed as brachial artery flow-mediated dilation using vascular ultrasound

SECONDARY OUTCOMES:
Nitroglycerin-mediated dilation | 4 weeks
  Non-endothelium-dependent dilation will be assessed by measuring the dilator response to sublingual nitroglycerin using vascular ultrasound
Carotid-Femoral Pulse Wave Velocity | 4 weeks
  Central aortic stiffness will be assessed as carotid-femoral pulse wave velocity using applanation tonometry
Reactive hyperemia | 4 weeks
  We will use vascular ultrasound to determine maximal hyperemic flow velocity in the brachial artery induced by 4-minute cuff occlusion.

OTHER OUTCOMES:
Fasting glucose and insulin | 4 weeks
  Fasting glucose and insulin

CONTACTS AND LOCATIONS:
Overall Officials: Robert E Eberhardt, MD, Principal Investigator — Boston University
Locations (1):
- Boston University School of Medicine, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No